CLINICAL TRIAL: NCT00746460
Title: The Effectiveness of CVD Risk Profiles When Used by Allied Health Care Providers (HCP) Within a "Groupe de Médecine de Famille": The Healthy Options Feasibility Study.
Brief Title: The Healthy Options Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Steven Grover, MD, Medical Director McGill Comprehensive Health Improvement Program, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLIN-08001
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Sedentary Lifestyle; Dyslipidemia; Hypertension; Cigarette Smoking; Diabetes
Keywords: primary prevention; patient knowledge; nurse; exercise; smoking cessation; weight loss
MeSH Terms: conditions — Obesity; Sedentary Behavior; Dyslipidemias; Hypertension; Cigarette Smoking; Diabetes Mellitus; Motor Activity; Smoking Cessation; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Behavioral
  Interventions: Behavioral: CVD risk profile

INTERVENTIONS:
Behavioral: CVD risk profile — Cardiovascular risk assessment and behavioral counselling

SUMMARY:
The investigators hypothesize that having health care providers other than physicians within a "Groupe de Médecine de Famille" conduct cardiovascular risk assessments and teach lifestyle interventions to primary prevention patients will increase the likelihood that patients will adopt and maintain healthy lifestyles. These objectives will be supported by providing subjects with a cardiovascular risk profile estimating the subject's risk of cardiovascular disease and teaching them how to use the resources related to lifestyle changes available on the www.myhealthcheckup.com Web site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 30-79 years of age without known cardiovascular disease but with one or more risk factors such as obesity, a sedentary lifestyle, dyslipidemia, hypertension, cigarette smoking, or diabetes
* Have provided informed consent
* Recent (past 6 months) fasting lipid profile results in the medical charts

Exclusion Criteria:

* Unable or unlikely to follow and/or complete study or evidence of uncooperative attitude
* Subject is not literate in either French or English
* Subject does not have easy and regular access to the Internet
* Exercise or weight loss are contra-indicated for medical reasons

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of using health care providers other than physicians within a GMF to conduct a CV risk assessment and intervention on primary prevention patients | 10 months

SECONDARY OUTCOMES:
Patient's CV risk factors and overall CV risk | 16 weeks
Subject's adherence with lifestyle changes and prescribed medications | 16 weeks
Satisfaction of the nurse | 10 months
Satisfaction of the patient | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grover, MD, Principal Investigator — McGill Cardiovascualr Health Improvement Program
Locations (1):
- McGill Cardiovascular Health Improvement Program, Montreal, Quebec, Canada

REFERENCES:
- See also: Web site used by study participants — http://www.myhealthcheckup.com